CLINICAL TRIAL: NCT04136002
Title: Evaluation of the ctDNA LUNAR Test in an Average Patient Screening Episode
Acronym: ECLIPSE
Status: Completed | Type: Observational
Sponsor: Guardant Health, Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Other Study IDs: 02-GI-002
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens will be retained in order to investigate the performance characteristics of the LUNAR-2 device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The ECLIPSE (Evaluation of the ctDNA LUNAR test in an Average Patient Screening Episode) study is a prospective, observational multi-site study without randomization. The primary objective of the study is to evaluate the performance characteristics of a blood-based ctDNA LUNAR-2 test to detect colorectal cancer in a screen-relevant, average risk population.

DETAILED DESCRIPTION:
The LUNAR-2 test has been developed to detect malignant disease in screen-relevant patients who would otherwise undergo screening for malignant disease using invasive methodologies such as colonoscopy. The intended use of such a test would be to return a result of ctDNA detected/ ctDNA not detected in a patient eligible for average risk screening for colorectal cancer. Those patients who receive a ctDNA detected result should undergo further investigation with colonoscopy.

In order to define the performance characteristics of the test in a relevant population, this study will perform a blood draw prior to the patient undergoing the standard of care colonoscopy (and all associated preparatory medications) and retrospectively compare the performance characteristics of the LUNAR-2 test with the findings of the index colonoscopy.

Outcomes of patients at one and two-years post-procedure will be collected as secondary endpoints to investigate the possibility of incidental, non-colorectal cancer cases and interval cancers that had not reached the clinical threshold for detection at the time of the index colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 45-84 years at time of consent
2. Intended to undergo screening colonoscopy
3. Considered by a physician or healthcare provider as being of 'average risk' for CRC
4. Willing to consent to blood draw pre-bowel preparation administration prior to undergoing colonoscopy within 60 days of the date of the investigational blood draw
5. Willing to consent to follow-up for two years as per protocol

Exclusion Criteria:

1. Undergoing colonoscopy for investigation of symptoms
2. Has undergone colonoscopy within preceding 9 years
3. Positive FIT/FOBT result within the previous 6 months
4. Has completed Cologuard or Epi proColon testing within the previous 3 years
5. History of colorectal cancer
6. History of any malignancy (patients who have undergone surgical removal of skin squamous cell cancer may be enrolled provided the procedure was completed at least 12 months prior to the date of provision of informed consent for the study)
7. Known diagnosis of inflammatory bowel disease
8. Currently taking any anti-neoplastic or disease-modifying anti-rheumatic drugs (DMARDs)
9. Positive family history of colorectal cancer, defined as having one or more first- degree relatives (parent, sibling, or child) with CRC at any age
10. Known hereditary/germline risk of colorectal cancer (for example, Lynch syndrome or Hereditary Non-Polyposis CRC [HNPCC], or Familial Adenomatous Polyposis [FAP])
11. Any major physical trauma (e.g. disruption of tissue, surgery, organ transplant, blood product transfusion) within the 30 days leading up to the provision of informed consent
12. Known medical condition which, in the opinion of the investigator, should preclude enrollment into the study
13. Participation in a clinical research study in which an experimental medication has been administered or may be administered within the 30 days leading up to providing informed consent or may be administered through the time of colonoscopy

Ages: 45 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Single cohort of patients aged between 45 and 84, with no known high risk features, undergoing routine colorectal cancer screening as standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 44467 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Sensitivity of colorectal cancer detection | 60 days
  Sensitivity of colorectal cancer detection
Specificity of advanced neoplasia detection | 60 days
  Specificity of advanced neoplasia detection

SECONDARY OUTCOMES:
Positive predictive value of colorectal cancer detection | 60 days
  Positive predictive value of colorectal cancer detection
Negative predictive value of colorectal cancer detection | 60 days
  Negative predictive value of colorectal cancer detection
Sensitivity and specificity of advanced adenoma detection | 60 days
  Sensitivity and specificity of advanced adenoma detection

CONTACTS AND LOCATIONS:
Overall Officials: Craig Eagle, MD, Principal Investigator — Guardant Health, Inc.
Locations (270):
- United States (270):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Lakeview Clinical Research, Guntersville, Alabama
  - Medical Affiliated Research Center, Huntsville, Alabama
  - Jasper Summit Research LLC, Jasper, Alabama
  - Hope Research Institute, Chandler, Arizona
  - Southeast Valley Gastroenterology, Chandler, Arizona
  - Prime Medical Group, LLC, Gilbert, Arizona
  - Hope Research Institute, Glendale, Arizona
  - GI Research Associates, LLC, Phoenix, Arizona
  - "Forty-Third Medical Associates Absolute Clinical Research", Phoenix, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Novak Clinical Research, Tucson, Arizona
  - Del Sol Research Management, LLC, Tuscon, Arizona
  - Preferred Research Partners, Inc, Little Rock, Arkansas
  - Premier Gastroenterology, Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Associated Gastroenterology Medical Group, Anaheim, California
  - InSite Digestive Health Care, Arcadia, California
  - Gastroenterology, Burlingame, California
  - Ventura County Gastroenterology Medical Group, Camarillo, California
  - Hope Clinical Research, Canoga Park, California
  - Alliance Research Institute, Canoga Park, California
  - Gastro SB Clinic, Chula Vista, California
  - Precision Research Institute, Chula Vista, California
  - BG Clinical Research and affiliate of The Clinical Trials Network, LLC, Encinitas, California
  - Diagnamics, Inc, Encinitas, California
  - Helping Hands Healthcare Group, Fullerton, California
  - Paragon RX Clinical, Inc., Garden Grove, California
  - Digestive Health Research of Southern California, Huntington Beach, California
  - United Medical Doctors, Irvine, California
  - Gastro Care Institute, Lancaster, California
  - LA Gastroenterology Group, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - Gastroenterology Associates of Beverly Hills, Los Angeles, California
  - Knowledge Research Center, Orange, California
  - InSite Digestive Health Care-San Gabriel, Oxnard, California
  - Desert Oasis Healthcare Medical Group, Palm Springs, California
  - Palm Tree Clinical, Inc, Palm Springs, California
  - InSite Digestive Health Care - Gastroenterology Associates, Pasadena, California
  - Northern California Research, Sacramento, California
  - San Diego Gastroenterology Medical Associates, San Diego, California
  - SDG Clinical Research, Inc., San Diego, California
  - Precision Research Institute, San Diego, California
  - Medical Associates Research Group, San Diego, California
  - FOMAT Simoni AGI Medical, Thousand Oaks, California
  - Med Partners, Inc. dba Premiere Medical Center of Burbank, Inc, Toluca Lake, California
  - Curebase, Walnut Creek, California
  - Clinical Research of California, Walnut Creek, California
  - Gastroenterology Associates of Fairfield County, Bridgeport, Connecticut
  - CMR of Greater New Haven, LLC, Hamden, Connecticut
  - Yale University, New Haven, Connecticut
  - Innovative Medical Research of South Florida, Inc., Aventura, Florida
  - Reciomed Clinical Research Network, Inc., Boynton Beach, Florida
  - Clinical Research of South Florida, an AMR Company, Coral Gables, Florida
  - Dolphin Medical Research, Doral, Florida
  - University of Florida College of Medicine, Gainesville, Florida
  - Palmetto Research, LLC, Hialeah, Florida
  - The Center for Gastrointestinal Disorders, Hollywood, Florida
  - Research Centers of America, Hollywood, Florida
  - Health Awareness, Inc, Jupiter, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Multi-Specialty Research Associates, Lake City, Florida
  - University Clinical Research-DeLand, LLC dba Accel Research Sites, Lake Mary, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - University Clinical Research-DeLand, LLC dba Accel Research Sites, Melbourne, Florida
  - Crystal Biomedical Research, Miami Lakes, Florida
  - Ocala GI Research, LLC, Ocala, Florida
  - Sarkis Clinical Trials, Ocala, Florida
  - Gastroenterology of Greater Orlando, Orange City, Florida
  - Gastroenterology Institute of Orlando, Orlando, Florida
  - Advanced Gastroenterology Associates, LLC, Palm Harbor, Florida
  - Precision Clinical Research, LLC, Sunrise, Florida
  - Guardian Angel Research Center, LLC, Tampa, Florida
  - Digestive Health Care of Georgia, Atlanta, Georgia
  - Emory University School of Medicine, Atlanta, Georgia
  - Metro Atlanta Gastroenterology, LLC., Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Gastroenterology Consultants of Augusta, Evans, Georgia
  - SKY Clinical Research Network Group, Lawrenceville, Georgia
  - Infinite Clinical Trials, Riverdale, Georgia
  - WR-Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Rolphe Adult and Pediatric Medicine, Union City, Georgia
  - Christie Clinic, Champaign, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - Curebase, Chicago, Illinois
  - Digestive Health Services, Downers Grove, Illinois
  - Edward Hines Jr. VA Hospital, Hines, Illinois
  - Gastroenterology & Internal Medicine Specialist, SC, Avicenna Clinical Research, Lake Barrington, Illinois
  - Suburban Gastroenterology Ltd, Naperville, Illinois
  - Comprehensive Gastrointestinal Health, Northbrook, Illinois
  - DM Clinical Research, Oak Lawn, Illinois
  - Rockford Gastroenterology Associates, Ltd., Rockford, Illinois
  - Digestive Research Alliance of Michiana, South Bend, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Alliance for Multispecialty Research, LLC, El Dorado, Kansas
  - West Glen Gastrointestinal Consultants, P.A., Shawnee, Kansas
  - Alliance for Multispecialty Research-Wichita West, Wichita, Kansas
  - Kansas Gastroenterology, LLC, Wichita, Kansas
  - Tri-State Gastroenterology Associates, Crestview Hills, Kentucky
  - University of Louisville Research Foundation, Louisville, Kentucky
  - Robley Rex VA Medical Center, Louisville, Kentucky
  - Northlake Gastroenterology Associates, Covington, Louisiana
  - Northlake Gastroenterology Associates, Hammond, Louisiana
  - CroNola LLC, Houma, Louisiana
  - Gastroclinic, Lafayette, Louisiana
  - Clinical Trials of SWLA, LLC, Lake Charles, Louisiana
  - Delta Research Partners, Monroe, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Gastro Center of Maryland, Columbia, Maryland
  - Centennial Medical Group, Elkridge, Maryland
  - Frederick Gastroenterology Associates, Frederick, Maryland
  - Mid-Atlantic GI Research, Greenbelt, Maryland
  - Meridian Clinical Research, Rockville, Maryland
  - Digestive Health Specialists, Chelmsford, Massachusetts
  - South Suburban Gastroenterology, South Weymouth, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Onyx Clinical Research, Rochester Hills, Michigan
  - Covenant HealthCare, Saginaw, Michigan
  - Revive Research Institute, LLC, Southfield, Michigan
  - Clinical Research Institute of Michigan, LLC, Troy, Michigan
  - Curebase, Eagan, Minnesota
  - Gastroenterology Associates of Mississippi, Columbus, Mississippi
  - Southern Therapy and Advanced Research, Jackson, Mississippi
  - Quinn Healthcare, Ridgeland, Mississippi
  - Clinical Research Professionals, LLC, Chesterfield, Missouri
  - Digestive Health Specialists, LLC, Saint Joseph, Missouri
  - Saint Louis University GI & Hepatology Research Unit, St Louis, Missouri
  - Washington University School of Medicine Gastroenterology, St Louis, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Skyline Medical Center, PC/CCT Research, Elkhorn, Nebraska
  - Midwest Regional Health Services, LLC/CCT Research, Omaha, Nebraska
  - Excel Clinical Research, Las Vegas, Nevada
  - Wr-Crcn, Llc, Las Vegas, Nevada
  - Gastroenterology Consultants, Reno, Nevada
  - Advanced Research Institute, Reno, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Allied Health Clinical Research Organization, LLC, Brick, New Jersey
  - Gastroenterology Associates Of New Jersey, Clifton, New Jersey
  - AIG Digestive Disease Research, Florham Park, New Jersey
  - Allied Health Clinical Research Organization, LLC, Freehold, New Jersey
  - Hackensack Digestive Disease Associates, Hackensack, New Jersey
  - Digestive Healthcare Center, Hillsborough, New Jersey
  - Allied Health Clinical Research Organization, Jackson, New Jersey
  - Gastroenterology Associates Of New Jersey, Montclair, New Jersey
  - Dr. Howard N. Guss and Dr. Gagan Beri, Ocean City, New Jersey
  - Gastroenterology Associates Of New Jersey, Ridgewood, New Jersey
  - Teaneck Gastroenterology Associates, Teaneck, New Jersey
  - Advanced Gastroenterology Group, Union, New Jersey
  - Gastroenterology Associates Of New Jersey, Wayne, New Jersey
  - North Jersey Gastroenterology, Wayne, New Jersey
  - Gastroenterology Associates Of New Jersey, Woodland Park, New Jersey
  - Lovelace Scientific Resources, Inc., Albuquerque, New Mexico
  - Sam Moskowitz, MD, Brooklyn, New York
  - NY Scientific, Brooklyn, New York
  - Associated Gastroenterologists of Central New York, Camillus, Camillus, New York
  - Associated Gastroenterology of Central New York, East Syracuse, New York
  - Associated Gastroenterologists of Central New York, Fayetteville, New York
  - Intercity Gastroenterology, Fresh Meadows, New York
  - South Island Gastro, Lawrence, New York
  - East End Gastroenterology & Hepatology, Manorville, New York
  - Gastrointestinal Associates of Rockland, New City, New York
  - Smart Medical Research, Richmond Hill, New York
  - Syracuse Gastro Associates, Syracuse, New York
  - Digestive Disease Medicine Of Central New York, Utica, New York
  - GastroCare LI, Valley Stream, New York
  - Gastrointestinal Specs Lng Is, Wantagh, New York
  - Eric L. Tatar, MD, West Nyack, New York
  - Digestive Health Partners, Asheville, North Carolina
  - Cary Gastro Associates, Cary, North Carolina
  - UNC Division of Gastroenterology and Hepatology, Chapel Hill, North Carolina
  - Charlotte Gastroenterology & Hepatology, PLLC, Charlotte, North Carolina
  - Carolina Digestive Health Associates, PA, Charlotte, North Carolina
  - Javara Research, Charlotte, North Carolina
  - Carolinas Research Center, Charlotte, North Carolina
  - Carolina Digestive Health Associates, PA, Concord, North Carolina
  - Northeast GI Research Division, Concord, North Carolina
  - Coastal Research Institute, LLC, Fayetteville, North Carolina
  - Medication Management LLC, Greensboro, North Carolina
  - Pinehurst Medical Clinic, Pinehurst, North Carolina
  - Carolina's GI Research, LLC, Raleigh, North Carolina
  - PMG Research of Raleigh, Raleigh, North Carolina
  - Boice Willis Clinic, PA, Rocky Mount, North Carolina
  - PMG Research of Salisbury, LLC, Salisbury, North Carolina
  - Piedmont HealthCare, PA, Statesville, North Carolina
  - Wilmington Health, Wilmington, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - PMG Research of Winston, Winston-Salem, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - Plains Clinical Research Center, LLC, Fargo, North Dakota
  - Gastroenterology Associates of Cleveland, Beachwood, Ohio
  - Dayton Gastroenterology, Inc., Beavercreek, Ohio
  - Dayton Gastroenterology, Beavercreek, Ohio
  - Gastro Health Research, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - ClinOhio Research Services, Columbus, Ohio
  - Advance Clinical Research, Dayton, Ohio
  - META Medical Research Institute, Dayton, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - DSI Research, LLC, Springboro, Ohio
  - University of Toledo Internal Medicine Clinic, Toledo, Ohio
  - Avamar Gastroenterology and Center, Warren, Ohio
  - Northshore Gastroenterology & Endoscopy Center, Westlake, Ohio
  - Digestive Disease Specialists, Inc, Oklahoma City, Oklahoma
  - Options Health Research, LLC, Tulsa, Oklahoma
  - Fanno Creek Group, Portland, Oregon
  - The Oregon Clinic - Gastroenterology East, Portland, Oregon
  - Eastern Pennsylvania GI & Liver Specialists, Allentown, Pennsylvania
  - US Digestive Health at Blair, Altoona, Pennsylvania
  - Valley Gastroenterology Associates, Beaver Falls, Pennsylvania
  - Susquehanna Research Group, LLC, Camp Hill, Pennsylvania
  - Susquehanna Research Group, Harrisburg, Pennsylvania
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Einstein Medical Center Department of Digestive Disease and Transplantation, Philadelphia, Pennsylvania
  - Frontier Clinical Research, LLC, Uniontown, Pennsylvania
  - GIMED Associates, Inc., Cranston, Rhode Island
  - GIMED Associates, Inc., Narragansett, Rhode Island
  - Digestive Disease Research Center, Greenwood, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Southeast Medical Research/Elms Research, North Charleston, South Carolina
  - South Carolina Clinical Research LLC, Orangeburg, South Carolina
  - PPCP Division of Gastroenterology LLC, Summerville, South Carolina
  - Invocare Medical Research & Healthcare Center, West Columbia, South Carolina
  - Elligo Clinical Research Center, Austin, Tennessee
  - Erlanger Health Clinical Resarch, Chattanooga, Tennessee
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Gastro One, Germantown, Tennessee
  - Helios Clinical Research lLC, Jackson, Tennessee
  - The Jackson Clinic, PA, Jackson, Tennessee
  - The Jackson Clinic, Jackson, Tennessee
  - East Tennessee Research Institute, Johnson City, Tennessee
  - Tri-Cities Gastroenterology, Kingsport, Tennessee
  - Gastrointestinal Associates, P.C., Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Advanced Gastroenterology, Union City, Tennessee
  - Allied Digestive Disease Center, Cypress, Texas
  - Northside Gastroenterology Associates, Cypress, Texas
  - Uma Mohan MD PA, Cypress, Texas
  - El Paso Integrated Physicians Group, P.A., El Paso, Texas
  - Digestive Health Associates, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Biopharma Informatic, Houston, Texas
  - Diversified Medical Practices, Houston, Texas
  - Houston Digestive Diseases Consultants, Houston, Texas
  - Memorial Hermann Surgery Center, Houston, Texas
  - Protenium Clinical Research Inc., Hurst, Texas
  - Biopharma Informatic, McAllen, Texas
  - Gastroenterology Consultants, P.A., Pasadena, Texas
  - Clinical Associates in Research Therapeutics of America, San Antonio, Texas
  - Gastroenterology Partners of North Houston, Shenandoah, Texas
  - Texas Gastroenterology Associates/A1 Clinical Network, Spring, Texas
  - Gastroenterology Associates of Texas, PA, Sugar Land, Texas
  - Texas Gastro Consultants, Tomball, Texas
  - Digestive Health Research of North Texas, Wichita Falls, Texas
  - Progressive Clinical Research, Bountiful, Utah
  - Advanced Research Institute, Ogden, Utah
  - Advanced Research Institute Granite Peaks Gastroenterology, Sandy City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Verity Research, Fairfax, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - The Gastroenterology Group, Reston, Virginia
  - GI Select Health Research, LLC, Richmond, Virginia
  - Tidewater Physicians Multispecialty Group Clinical Research, Williamsburg, Virginia
  - Washington Gastroenterology, Bellevue, Washington
  - Western Washington Medical Group, Inc, Everett, Washington
  - Velocity Clinical Research, Spokane, Washington
  - Holy Family Memorial, Inc, Manitowoc, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - GI Associates, Stevens Point, Wisconsin
  - GI Associates, Wausau, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lo YMD. Cell-free DNA for Colorectal Cancer Screening. N Engl J Med. 2024 Mar 14;390(11):1047-1050. doi: 10.1056/NEJMe2311101. No abstract available. PMID 38477993
- [Derived] Chung DC, Gray DM 2nd, Singh H, Issaka RB, Raymond VM, Eagle C, Hu S, Chudova DI, Talasaz A, Greenson JK, Sinicrope FA, Gupta S, Grady WM. A Cell-free DNA Blood-Based Test for Colorectal Cancer Screening. N Engl J Med. 2024 Mar 14;390(11):973-983. doi: 10.1056/NEJMoa2304714. PMID 38477985